CLINICAL TRIAL: NCT07193238
Title: Application of an Ashridge Training Model-Based Ethics and Moral Course in Newly Graduated Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ashridge Training Model; FNEF202115 (Other Grant/Funding Number: Fudan University School of Nursing Research Fund); SYSZ2303 (Other Grant/Funding Number: Key Project of Medical Education, Shanghai Medical College of Fudan University)
Record Dates: First submitted 2025-09-12; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Professional Sense of Mission; Professional Benefit Perception; Humanistic Care Ability; Theoretical Knowledge and Practical Skills Performance; New Graduated Nurses; The Ethics and Moral Course
Keywords: Ashridge Training Model; ethics education; moral education; newly graduated nurses

STUDY DESIGN:
Intervention Model Description: The Ashridge training model, originating in 1986, was developed by a research project team at Ashridge Management College. It divides training activities into three stages: discrete stage, integration stage, and cumulative stage. This model places significant emphasis on both individual and organizational learning.
Who Masked: Participant
Masking Description: The intervention study employed a single-blind design, keeping subjects unaware of the specific interventions and whether they were assigned to the control or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group underwent a conventional one-year training for newly graduated nurses, initially consisting of centralized training by the hospital and nursing departments, covering regulations, laws, medical ethics, nursing professional spirit, specialized theory, and basic operational training. Upon entering their respective departments, one-on-one mentorship was provided by instructors, teaching basic nursing, specialized disease care, basic and specialized nursing operations, and nursing workflows. Theoretical knowledge was delivered through PPT lectures, while nursing skill training included demonstrations, explanations, and organized practice. Real-time guidance was provided during the learning process, with periodic assessments in theory and practice to ensure learning outcomes.
- Intervention group (Experimental): In addition to the same training as the control group, the intervention group received the Ethics and Moral Course based on the Ashridge training model, tailored for newly graduated nurses.
  Interventions: Other: The Ethics and Moral Course based on the Ashridge training model

INTERVENTIONS:
Other: The Ethics and Moral Course based on the Ashridge training model — Based on the three-stage characteristics of the Ashridge training model, the developed the content of this ethics course. (1) Discrete stage (within 3 months of employment): This stage aims to initially cultivate the professional identity of new nurses, stimulating humanistic awareness. It primarily involves self-study, supplemented by instructor supervision and implicit positive guidance. (2) Integrated stage (4-6 months of employment): This stage combines professional identity with actual work, enhancing humanistic care abilities in practice. It emphasizes mutual sharing between instructors and new nurses, utilizing diverse training methods to promote experience and reflection. (3) Cumulative stage (7-12 months of employment): This stage develops critical thinking and ethical problem-solving abilities. It focuses on assessing comprehensive abilities in complex nursing situations, providing feedback on the teaching plan, and evaluating training effectiveness.
  Arms: Intervention group

SUMMARY:
The objective of this historical control trial is to evaluate the effectiveness of an Ethics and Moral Course, based on the Ashridge training model, in newly graduated nurses. The primary questions it aims to address are: (1) What is the impact of integrating moral education into the standardized training of newly employed nurses on their professional outlook? (2) Can this study enhance the humanistic care abilities and overall competencies of newly graduated nurses?

Researchers compared two groups of newly employed nurses (without work experience) at a specific hospital. The control group received conventional training, while the intervention group underwent a moral education curriculum designed in three stages based on the Ashridge training model, in addition to traditional training. Post-training, the two groups were compared in terms of their sense of professional mission, perceived professional benefits, humanistic care abilities, theoretical knowledge, and practical skills performance.

DETAILED DESCRIPTION:
With the continuous development of the healthcare sector, nursing personnel face increasingly higher professional demands. Newly graduated nurses, lacking work experience, are particularly prone to ethical dilemmas during their transition from nursing students to clinical practitioners. Ophthalmology and otolaryngology diseases often affect patients' sensory functions and quality of life, imposing higher competency requirements on Eye, Ear, Nose, and Throat (EENT) nurses. Standardized training, as a crucial transitional period for new nurses, presents an optimal opportunity to integrate ethical education, thereby fostering their professional outlook and moral qualities.

This study underscores the importance of structured ethical and moral education during this critical transition period. The investigators first developed an ethics and morality curriculum tailored for new EENT nurses based on the Ashridge training model, followed by a non-randomized controlled trial to evaluate its effectiveness. Newly employed nurses (new graduates without work experience) at a tertiary specialized hospital in Shanghai were selected as study subjects. Sixty new nurses employed between January 2022 and December 2022 served as the control group and received conventional training. Between January 2023 and December 2023, sixty newly employed nurses served as the intervention group, receiving an ethics and morality curriculum designed in three phases based on the Ashridge training model, in addition to conventional training.

A mixed-methods research design was adopted. The investigators surveyed the sense of professional mission, professional benefit perception, humanistic care ability, theoretical knowledge, practical skills, and scenario-based case simulation performance in both groups post-training. The qualitative component used purposive sampling to conduct semi-structured interviews with 18 new nurses. Thematic framework analysis was employed to extract viewpoints, categorize reasoning, and summarize themes.

The results indicated that the intervention group outperformed the control group across all measured parameters (P < 0.05). The results highlight the effectiveness of our course in enhancing the professional identity, ethical decision-making, and humanistic care abilities of newly graduated nurses. Our qualitative interviews further complemented the quantitative findings, providing valuable insights for the development of ethical and moral education courses for new nurses.

ELIGIBILITY:
Inclusion Criteria:

* Newly graduated nurses with no prior clinical nursing experience.
* Possession of a nurse licensure certificate.
* Currently undergoing a one-year standardized training for newly graduated nurses.
* Voluntary participation in the study with informed consent signed by the nurse.

Exclusion Criteria:

* Newly graduated nurses on medical leave exceeding three months or those in a non-working status during the study period, including maternity leave, sick leave, or vacation.
* Nurses with a recent history of major traumatic events leading to mental debilitation or psychological trauma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Professional Calling | Within 7 days after the completion of the training program
  Evaluation was conducted using the Professional Calling Scale. This scale consists of 12 items and is a unidimensional scale. It uses a Likert 5-point scale, ranging from 1 (strongly disagree) to 5 (strongly agree), resulting in a total score range of 12 to 60, with higher scores indicating a stronger sense of professional calling.
Professional Benefits | Within 7 days after the completion of the training program
  Evaluation was conducted using the Nurse Professional Benefits Scale. This scale comprises 29 items across five dimensions: Positive Professional Perception (5 items), Family and Friends' Recognition (7 items), Team Belongingness (5 items), Good Nurse-Patient Relationship (6 items), and Personal Growth (6 items). It uses a Likert 5-point scale, ranging from 1 (strongly disagree) to 5 (strongly agree), with a total score range of 29 to 145. Higher scores indicate a higher level of professional benefits for nurses.
Humanistic Caring Ability | Within 7 days after the completion of the training program
  Evaluation was conducted using the Nursing Students' Humanistic Caring Ability Scale. This scale consists of 45 items across eight dimensions: Instilling Beliefs and Hope (9 items), Humanitarian Altruistic Values (6 items), Health Education (7 items), Promoting Emotional Communication (5 items), Scientifically Solving Health Problems (4 items), Assisting in Meeting Basic Needs (4 items), Helping Solve to Difficulties (5 items), and Providing a Good Environment (5 items). It uses a Likert 5-point scale, with positive items scored from 4 (completely agree) to 0 (completely disagree), and 10 reverse-scored items from 0 (completely agree) to 4 (completely disagree), providing a total score range of 0 to 180. Higher scores indicate stronger humanistic caring abilities.

SECONDARY OUTCOMES:
Theoretical Knowledge and Practical Skills, and Scenario Simulation Exam Scores | During the last seven days of the training program
  Two groups of newly graduated nurses were assessed on fundamental nursing theory, practical nursing skills, and scenario-based case examinations. Standardized patients were portrayed by three nurses who had undergone rigorous standardized training and passed competency evaluations. The scenario-based case examinations included assessments of ophthalmology and otolaryngology workflows, evaluating the new nurses' abilities in nurse-patient communication, clinical judgment, emergency response, and practical skills.
Qualitative Research | Within 7 days after the completion of the training program
  A semi-structured interview method was used to gain in-depth insights into their perceptions of the Ethics and Moral Course, thereby complementing the quantitative research.

CONTACTS AND LOCATIONS:
Locations (1):
- EYE & ENT Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang Y. An Empirical Study on Evaluation of Humanistic Caring Ability of Nursing Undergraduates. Master, Fujian Medical University, 2007.
- [Background] Hu J. Study on Conceptual Framework and Evaluation Tool of Nurse's Perceived Professional Benefits. Master, Second Military Medical University, 2013.
- [Background] Dobrow SR and Tosti-Kharas J. Calling: The development of a scale measure. Personnel Psychology 2011; 64: 1001-1049.
- [Background] Zhou Y. Research on the Relationship between Career Calling, Career Commitment and Career Success. Master, Jilin University, 2013.
- [Background] Missen K, McKenna L, Beauchamp A. Satisfaction of newly graduated nurses enrolled in transition-to-practice programmes in their first year of employment: a systematic review. J Adv Nurs. 2014 Nov;70(11):2419-33. doi: 10.1111/jan.12464. Epub 2014 Jul 2. PMID 24989716
- [Background] Cavanagh N, Cockett G, Heinrich C, Doig L, Fiest K, Guichon JR, Page S, Mitchell I, Doig CJ. Compassion fatigue in healthcare providers: A systematic review and meta-analysis. Nurs Ethics. 2020 May;27(3):639-665. doi: 10.1177/0969733019889400. Epub 2019 Dec 12. PMID 31829113
- [Background] Reebals C, Wood T, Markaki A. Transition to Practice for New Nurse Graduates: Barriers and Mitigating Strategies. West J Nurs Res. 2022 Apr;44(4):416-429. doi: 10.1177/0193945921997925. Epub 2021 Mar 16. PMID 33724088
- [Background] Hallaran AJ, Edge DS, Almost J, Tregunno D. New Nurses' Perceptions on Transition to Practice: A Thematic Analysis. Can J Nurs Res. 2023 Mar;55(1):126-136. doi: 10.1177/08445621221074872. Epub 2022 Jan 24. PMID 35068206
- [Background] Rattanasirivilai P, Shirodkar AL. A study of the role and educational needs of ophthalmic specialist nurses. Br J Nurs. 2021 Jul 22;30(14):858-864. doi: 10.12968/bjon.2021.30.14.858. PMID 34288742
- [Background] Haahr A, Norlyk A, Martinsen B, Dreyer P. Nurses experiences of ethical dilemmas: A review. Nurs Ethics. 2020 Feb;27(1):258-272. doi: 10.1177/0969733019832941. Epub 2019 Apr 11. PMID 30975034